CLINICAL TRIAL: NCT06910449
Title: Hemithoracic Volumetric Modulated Arc Radiotherapy as Part of Lung-Sparing Multimodality Therapy in Patients With Malignant Pleural Mesothelioma Phase II Trial
Brief Title: Hemithoracic Arc Radiotherapy Post Pleural Decortication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Gamal, Assistant Lecturer of Radiation Oncology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RO2405-291-047-193
Record Dates: First submitted 2024-12-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm receiving postoperative radiotherapy (Experimental): single arm receiving post operative Radiotherapy to the hemithorax
  Interventions: Radiation: hemithoracic Volumetric Arc Radiotherapy post Pleural decortication

INTERVENTIONS:
Radiation: hemithoracic Volumetric Arc Radiotherapy post Pleural decortication — post operative delivery of hemithoracic Volumetric Arc Radiotherapy

SUMMARY:
Malignant Pleural Mesothelioma is an aggressive and refractory disease , the most aggressive treatment plan offered to these patients include trimodalitiy approach with chemotherapy as the mainstay of treatment . the rationale of post operative Radiotherapy is to sterilize the post operative volume to reduce local failure meanwhile minimizing toxicities in this trial we are going to assess the safety and efficacy of Radiotherapy in Mesothelioma patients poat Pleural decortication

DETAILED DESCRIPTION:
This study will include malignant Pleural Mesothelioma patients treated by trimodalitiy approach starting with neoadjuvant chemotherapy followed by surgery in the form of Pleural decortication then all patients will receive post operative hemithoracic radiation

ELIGIBILITY:
Inclusion Criteria:

* Evidence of metastatic disease.
* Underwent Pleural decortication.
* Able to provide informed consent.

Exclusion Criteria:

* Poor pulmonary function tests.
* Recurrent or palliative cases.
* Inability to attend full course of Radiotherapy or follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Acute Radiation Toxicity | weekly assessment during radiation course and monthly follow up for the first 6 months
  Questionnaire based Follow up about acute Radiation toxicity according to RTOG including dysnea , cough , chest pain , dysnea on effort from grade 1-5
late radiation toxicity | Bi-monthly fashion of minimum 6 months post radiation course
  follow up of patients using both Questionnaire and performing pulmonary function tests and Echo , focusing on DLCO & FEV1

CONTACTS AND LOCATIONS:
Locations (1):
- national Cancer Institute Cairo university, Cairo, Fom Elkhalig, Egypt

IPD SHARING:
Plan to Share IPD: No